CLINICAL TRIAL: NCT00674986
Title: A Clinical Study to Evaluate the Use of Episodic, Intensive Blood Glucose Monitoring in Persons With Non-insulin Treated Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000590; RDC-MI&A-01-2007
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Active Control Group (ACG) (Other): Participants in the Active Control Group received enhanced standard of care (more frequent clinic visits, free blood glucose meters and strips and point-of-care Hemoglobin A1c (HbA1c) test) for management of their Type 2 diabetes.
  Interventions: Device: Accu-Chek Aviva Glucose Meter
- Structured Testing Group (STG) (Experimental): Participants in the Structured Testing Group in addition to enhanced standard of care for the treatment of their Type 2 diabetes used the ACCU-CHEK® 360° View blood glucose analysis system (Tool) to monitor glucose levels at least quarterly.
  Interventions: Device: Accu-Chek 360° View Blood Glucose Analysis Tool; Device: Accu-Chek Aviva Glucose Meter

INTERVENTIONS:
Device: Accu-Chek 360° View Blood Glucose Analysis Tool
  Arms: Structured Testing Group (STG)
Device: Accu-Chek Aviva Glucose Meter

SUMMARY:
This randomized, parallel group study will determine whether the use of episodic, intensive glucose monitoring via the Accu-Chek 360 view blood glucose analysis system has a positive effect on overall glycemic control. Patients will be randomized into either the 'usual care' group, or the 'interventional group' supplemented with the Accu-Chek 360 view blood glucose analysis system. The effect of each treatment regimen on glycemic control will be assessed by measurement of change in baseline HbA1c values at 12 months. The anticipated time on study treatment is 1 year, and the target sample size is 504 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 25 years of age
* Type 2 diabetes for >= 1 year
* Hemoglobin A1c >= 7.5% and <=11%
* Diabetes managed by exercise and diet, prescription oral medication or an injectable incretin mimetic

Exclusion Criteria:

* Type 1 diabetes
* On any type of insulin therapy at start of study

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Petersen, Study Director — Roche Diagnostics GmbH
Locations (25):
- United States (25):
  - Mobile, Alabama
  - Pell City, Alabama
  - Chipley, Florida
  - Marianna, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - O'Fallon, Illinois
  - Fishers, Indiana
  - Indianapolis, Indiana
  - Flint, Michigan
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Cuyahoga Falls, Ohio
  - Zanesville, Ohio
  - Pottstown, Pennsylvania
  - High Point, South Carolina
  - Lancaster, South Carolina
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Crossville, Tennessee
  - Abingdon, Virginia

REFERENCES:
- [Derived] Fisher L, Polonsky W, Parkin CG, Jelsovsky Z, Amstutz L, Wagner RS. The impact of blood glucose monitoring on depression and distress in insulin-naive patients with type 2 diabetes. Curr Med Res Opin. 2011 Nov;27 Suppl 3:39-46. doi: 10.1185/03007995.2011.619176. Epub 2011 Sep 14. PMID 21916532
- [Derived] Polonsky WH, Fisher L, Schikman CH, Hinnen DA, Parkin CG, Jelsovsky Z, Petersen B, Schweitzer M, Wagner RS. Structured self-monitoring of blood glucose significantly reduces A1C levels in poorly controlled, noninsulin-treated type 2 diabetes: results from the Structured Testing Program study. Diabetes Care. 2011 Feb;34(2):262-7. doi: 10.2337/dc10-1732. PMID 21270183
- [Derived] Polonsky W, Fisher L, Schikman C, Hinnen D, Parkin C, Jelsovsky Z, Amstutz L, Schweitzer M, Wagner R. The value of episodic, intensive blood glucose monitoring in non-insulin treated persons with Type 2 Diabetes: design of the Structured Testing Program (STeP) study, a cluster-randomised, clinical trial [NCT00674986]. BMC Fam Pract. 2010 May 18;11:37. doi: 10.1186/1471-2296-11-37. PMID 20482765

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 770 patients were screened. 522 patients were enrolled in the study. 23 patients at 1 site used the incorrect self monitored blood glucose device and were excluded. 499 patients met inclusion/exclusion criteria and were included in the analyses.
Period: Overall Study
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Started | 230 | 269
Intent to Treat Population | 227 | 256
Completed | 187 | 188
Not Completed | 43 | 81
Not completed — Adverse Event | 2 | 1
Not completed — Subject withdrew consent | 12 | 19
Not completed — Lost to Follow-up | 25 | 53
Not completed — Other reasons | 4 | 8

BASELINE CHARACTERISTICS:
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG) | Total
Number analyzed (Participants) | 227 | 256 | 483
Age Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.2) | 54.8 (10.1) | 55.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 121 | 226
  Male | 122 | 135 | 257

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at Month 12
Description: Blood was collected at Baseline and Month 12 and analyzed at a central laboratory for HbA1c. Results were calculated using a Linear Mixed Model with study group, visit, group-by-visit interaction, baseline HbA1c, gender, age, and race as fixed effects; and site and subject as random effects. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Month 12
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 227 | 256
Percent | -0.88 (0.10) | -1.16 (0.09)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p = 0.0416, Fisher Exact; Difference = 0.28, 95% CI 2-sided [0.01 to 0.54], Standard Error of Mean 0.14

2. Secondary Outcome: Number of Visits With Diabetic Medication and/or Lifestyle Change Recommendations
Description: Treatment intensification was assessed at each clinic visit. The physician evaluated the patient and made recommendations of a change in two areas: changes in diabetic medication and/or changes in lifestyle (such as diet, exercise and education.)
Time Frame: 12 Months
Population: Intent to treat population included all enrolled participants who completed the Baseline training visit. Participants who dropped out before Month 1 visit were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 218 | 237
Visits | 1.1 (1.0) | 2.7 (1.5)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p < 0.0001, Fisher Exact

3. Secondary Outcome: Change From Baseline in Depression Severity (PHQ-8)
Description: The Patient Health Questionnaire-8 (PHQ-8) is an eight-item patient questionnaire to measure the severity of depression disorders over the previous 2 weeks. Each item is rated on a 4-point scale of: 0=not at all to 3=nearly every day. The total score for all items range from 0 (best) to 24 (worst). Results were calculated using a Linear Mixed Model with study group, visit, group-by-visit interaction, baseline PHQ-8, gender, age, and race as fixed effects; and site and subject as random effects. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Month 12
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 227 | 256
Score on a scale | -1.1 (0.3) | -1.7 (0.3)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p = 0.2777, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in the Diabetes Distress Scale (DDS)
Description: Participants rated their level of diabetes distress by answering 17 questions in in the following areas: Regimen-related Distress, Emotional Burden, Diabetes-related Interpersonal Distress and Physician-related Distress (PD) on a 6-point scale: 1=Not a problem to 6=A very serious problem. The Average Total score ranged from 1 (best) to 6 (worst). Results were calculated using a Linear Mixed Model with study group, visit, group-by-visit interaction, baseline DDS, gender, age, and race as fixed effects; and site and subject as random effects. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Month 12
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 227 | 256
Score on a scale | -0.40 (0.07) | -0.55 (0.06)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p = 0.1160, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in the World Health Organization (WHO-5) Well-being Index
Description: Participants used the WHO-5 to rate their well-being (feeling good and cheerful) for the past 2 weeks using a 6-point scale: 0=At no time to 5=All of the time for a total possible score of 0 (worst) to 100 (best). Results were calculated using a Linear Mixed Model with study group, visit, group-by-visit interaction, baseline WHO-5, gender, age, and race as fixed effects; and site and subject as random effects. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Month 12
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 227 | 256
Score on a scale | 4.1 (1.5) | 7.4 (1.5)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p = 0.1146, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in Confidence in Diabetes Self-Care (CIDS-2)
Description: Participants rated how confident they felt about managing each of 20 diabetes self-care tasks using the CIDS-2 questionnaire. Responses were given on a 5-point scale ranging from 1=not at all confident to 5=completely confident for a total possible score of 20 (worst) to 100 (best). Results were calculated using a Linear Mixed Model with study group, visit, group-by-visit interaction, baseline CIDS-2, gender, age, and race as fixed effects; and site and subject as random effects. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Month 12
Population: Per protocol population included all enrolled participants who completed the baseline training visit, completed at least 4 of 5 clinical visits, and had evaluable HbA1c data at Month 12. The Structured Testing Group also had to have at least 80% of the blood glucose values.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 161 | 130
Score on a scale | 2.7 (1.1) | 5.8 (1.1)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p = 0.0470, t-test, 2 sided

7. Secondary Outcome: Mean Number of Subject Monitored Blood Glucose (SMBG) Tests Per Day
Description: SMBG data for all participants was collected by the glucose meter and were uploaded directly to a web server. The mean number of SMBG tests/day was calculated for the entire study period.
Time Frame: 12 Months
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Measure: Least Squares Mean (Standard Error); unit: Tests/day
Arm/Group | Active Control Group (ACG) | Structured Testing Group (STG)
Number analyzed (Participants) | 227 | 256
Tests/day | 1.15 (0.80) | 0.89 (0.70)
Statistical Analysis 1: Comparison: Active Control Group (ACG) vs Structured Testing Group (STG); Test type: Superiority or Other; p = 0.0003, t-test, 2 sided

8. Secondary Outcome: Glycemic Variability Pre and Post-Prandial Excursions at Each Meal
Description: Glycemic Variability was evaluated in the STG group for each 3-day set that corresponded to the days the subjects completed the tool before each post-baseline clinic visit. Some parameters used to estimate glycemic variability over the 3-day profile included mean and maximum post-prandial glucose excursions (differences between pre- and post-meal blood glucose levels), mean blood glucose and mean amplitude of glycemic excursion.
  The calculation used a Linear mixed model with visit, Month 1 value, gender, age and race (White and Non-White) as fixed effects; and site and subject as random effects.
Time Frame: Month 1, Month 12
Population: Intent to treat population included all enrolled participants who completed the baseline training visit.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Structured Testing Group (STG)
Number analyzed (Participants) | 256
mg/dL
  Post-Prandial Glucose Excursion Breakfast Month 1 | 44.0 (2.3)
  Post-Prandial Glucose ExcursionBreakfast Month 12 | 34.7 (2.7)
  Post-Prandial Glucose Excursion Lunch Month 1 | 25.0 (2.4)
  Post- Prandial Glucose Excursion Lunch Month 12 | 17.3 (2.8)
  Post-Prandial Glucose Excursion Supper Month 1 | 33.6 (2.8)
  Post-Prandial Glucose Excursion Supper: Month 12 | 25.8 (3.3)
  Mean Amplitude of Glucose Excursions: Month 1 | 38.5 (0.9)
  Mean Amplitude of Glucose Excursions: Month 12 | 34.3 (1.0)
  Maximum Glucose Rise: Breakfast Month 1 | 80.2 (2.9)
  Maximum Glucose Rise: Breakfast Month 12 | 64.0 (3.5)
  Maximum Glucose Rise: Lunch Month 1 | 65.6 (3.2)
  Maximum Glucose Rise: Lunch Month 12 | 53.3 (3.8)
  Maximum Glucose Rise: Supper Month 1 | 72.3 (3.5)
  Maximum Glucose Rise: Supper Month 12 | 60.8 (4.1)

ADVERSE EVENTS:
Arm/Group | Structured Testing Group (STG) | Active Control Group (ACG)
Serious Adverse Events (participants affected / at risk) | 14/256 | 21/227
Other Adverse Events (participants affected / at risk) | 33/256 | 35/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Structured Testing Group (STG) (N=256) | Active Control Group (ACG) (N=227)
Atrial fibrillation (Cardiac disorders) | 0 | 2
SVT (Supraventricular tachycardia) (Cardiac disorders) | 0 | 1
Atrial fibrillation/bradycardia (Cardiac disorders) | 0 | 1
Exacerbation of coronary artery disease (Cardiac disorders) | 0 | 1
Emergency CABG x 5 (Coronary artery bypass graft) (Cardiac disorders) | 0 | 1
Artherosclerotic coronary disease (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Blockage in left descending coronary artery (Cardiac disorders) | 1 | 0
MVA - high speed (Motor vehicle accident) (Injury, poisoning and procedural complications) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Abdominal pain (General disorders) | 0 | 1
Mid sternal chest pain, acute onset (General disorders) | 1 | 0
Chest pain associated with pulled muscle (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Anterior and epigastric chest pain (General disorders) | 0 | 1
Acute cholecystitus (Hepatobiliary disorders) | 0 | 1
Biliary pancreatitis (Hepatobiliary disorders) | 0 | 1
Acute bronchitis (Infections and infestations) | 0 | 1
Pneumonia/bronchitis (Infections and infestations) | 0 | 1
Influenza a (Infections and infestations) | 0 | 1
Arm and leg swelling (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Intractable pain status post lumbar fusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Recurrent colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Left breast mastectomy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign tumor on thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vertigo/labyrinthitis/ataxia (Nervous system disorders) | 0 | 1
Brain stem CVA (Cerebrovascular accident) (Nervous system disorders) | 0 | 1
Major depressive symptoms - emptiness, nervousness (Psychiatric disorders) | 1 | 0
Major depressive disorder, recurrent, severe and adjustment disorder (Psychiatric disorders) | 1 | 0
Complex fluid collection posterior to the operative site (Injury, poisoning and procedural complications) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Congestive heart failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Worsening chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cellulitis of leg, left lower extremity (Skin and subcutaneous tissue disorders) | 1 | 0
Blister on right foot big toe (Skin and subcutaneous tissue disorders) | 1 | 0
Feeding tube placed problems eating (Surgical and medical procedures) | 0 | 1
Lower lumbar surgery (Surgical and medical procedures) | 0 | 1
Lower lumber decompression & laminectomy at L3-4, lumbar decompression, laminectomy, fusion at L4-5 (Surgical and medical procedures) | 0 | 1
Possible RIND (Reversible ischemic neurologic deficit) (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Structured Testing Group (STG) (N=256) | Active Control Group (ACG) (N=227)
Upper respiratory tract infection (Infections and infestations) | 18 | 20
Sinusitis (Infections and infestations) | 15 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.